CLINICAL TRIAL: NCT03942692
Title: What is the Allergy Follow-up for Children After Anaphylactic Reaction? AFCAR : Allergy Follow-up for Children After Anaphylactic Reaction
Acronym: SAPRA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0493
Record Dates: First submitted 2019-05-07; First posted 2019-05-08 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Anaphylaxis; Allergic Reaction
MeSH Terms: conditions — Anaphylaxis; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with anaphylactic reaction: Children who underwent an anaphylactic reaction between the 1st July 2014 and the 31st June 2016 treated in Paediatric Emergency Department of Femme-Mère-Enfant Hospital in Lyon in France.
  Interventions: Other: Phone call questionnaire

INTERVENTIONS:
Other: Phone call questionnaire — Questionnaire for parents of subject about :
  * the frequency of consultations with an allergist
  * the information of the general practitioner or pediatrician
  * the prescription of epinephrin auto-injector
  * the frequency of renewal of epinephrin auto-injector
  * the specialty of doctor who prescribed the renewal
  * the implementation of specific measures in schools
  * the frequency of renewal of specific measures in schools
  * the number of recurrence of anaphylactic reaction
  * the use of medical advice in case of recurrence of anaphylactic reaction

SUMMARY:
Anaphylaxis is an allergic reaction potentially fatal. The treatment is based on injection of epinephrin as soon as possible. Guidelines by the World Allergic Organisation highlight the importance of medical follow-up. This follow-up consists of an allergy consultation, the prescription and demonstration of epinephrin auto-injector and the implementation of specific measures in schools. There is no study about the recurrence of anaphylactic reaction outside the hospital.

The purpose of this study is to evaluate the allergy follow-up of children after anaphylactic reaction. The secondary objective is to evaluate the use of medical advice in case of recurrence of anaphylactic reaction.

Investigators will use a phone call questionnaire for parents of children who underwent an anaphylactic reaction between the 1st July 2014 and the 31st June 2016 treated in the Paediatric Emergency Department in Femme-Mère-Enfant Hospital in Lyon in France. 179 children could be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age from 0 to 17
* Anaphylactic reaction meeting the criteria of Sampson et al. treated in Paediatric Emergency Department of Femme-Mère-Enfant Hospital in Lyon in France
* Anaphylactic reaction treated between the 1st July 2014 and the 31st June 2016

Exclusion Criteria:

- No agreement from patient or parents to participate in the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children from 0 to 18 year old who underwent an anaphylactic reaction between the 1st July 2014 and the 31st June 2016 treated in Paediatric Emergency Department of Femme-Mère-Enfant Hospital in Lyon in France.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Allergy follow-up | About 15 minutes
  Allergy follow-up evaluation with :
  * the frequency of consultations with an allergist
  * the information of the general practitioner or pediatrician
  * the prescription of epinephrin auto-injector
  * the frequency of renewal of epinephrin auto-injector
  * the specialty of doctor who prescribed the renewal
  * the implementation of specific measures in schools
  * the frequency of renewal of specific measures in schools
  * the number of recurrence of anaphylactic reaction
  * the use of medical advice in case of recurrence of anaphylactic reaction

CONTACTS AND LOCATIONS:
Locations (1):
- Paediatric Emergency Department in Femme-Mère-Enfant Hospital, Bron, France